CLINICAL TRIAL: NCT06937658
Title: Remote Alert Pathway To Optimize CaRe of Cardiac Implantable Electrical Devices
Acronym: RAPTOR-CIED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Daniel B. Kramer, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLACER-2023C3-34968
Record Dates: First submitted 2025-04-08; First posted 2025-04-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pacemaker DDD; Implantable Defibrillator User

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Guideline-based Care (Active Comparator): Remote monitoring programming scheduled for alert transmissions, patient-initiated transmissions, and routine transmissions (scheduled to occur every 90 days from the date of enrollment in the study); in-office interrogations on at least an annual basis
  Interventions: Device: Guideline-based care
- Alert-based Care (Active Comparator): Remote monitoring programming scheduled for alert transmissions and patient-initiated transmissions only
  Interventions: Device: Alert-based care

INTERVENTIONS:
Device: Alert-based care — Alert-based care is an alternative strategy for longitudinal management of patients with wireless pacemakers and implantable defibrillators
  Arms: Alert-based Care
Device: Guideline-based care — Guideline-based care is the current typical standard for longitudinal management of patients with wireless pacemakers and implantable defibrillators
  Arms: Guideline-based Care

SUMMARY:
The Remote Alert Pathway to Optimize Care of Cardiac Implantable Electrical Devices (RAPTOR-CIED) Study is a pragmatic, multi-center, randomized trial with 1:1 patient-level randomization comparing the safety and effectiveness of alert-driven care versus guideline-based care for patients with wireless cardiac implantable electrical devices (CIEDs).

The study will be conducted in 2 phases: a Feasibility Phase and a Main Phase. This registration outlines the goals and design features of the Feasibility Phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged > 18 years
2. Clinically stable by investigator assessment
3. Has a newly implanted or existing wireless CIED: single, dual-chamber, biventricular, subcutaneous/extravascular, and leadless systems are all eligible, including pacemakers or implantable cardioverter-defibrillators (ICDs)
4. CIED is from one of the 4 major CIED manufacturers in the US market (99% of implants in the US): Medtronic, Boston Scientific, Abbott, Biotronik
5. Currently enrolled in remote monitoring as part of standard of care
6. Primary clinical electrophysiology follow-up at the enrolling center
7. Understands spoken and written English, Spanish, or Portuguese
8. Has sufficient cognitive function to answer standardized questions about study rationale and procedures.

Exclusion Criteria:

1. Presence of insertable cardiac monitor, either in isolation or in combination with any other CIED
2. Listed for cardiac transplantation prior to enrollment (N.B. if a patient becomes listed for transplantation during the study, they may continue study participation)
3. Participation in another study related to novel CIED technology or remote monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment | 6 months
  Number of patients enrolled and randomized per site and per month, and cumulatively
Adherence | 6 months
  Proportion of cross-over

SECONDARY OUTCOMES:
Major adverse cardiac events | 6 months
  Incidence of MACE (i.e., death, stroke or systemic embolism, and unplanned cardiac device procedure)
Major adverse cardiac events | 6 months
  Incidence of arrhythmia events, individual components of MACE, and health services use (i.e., hospital presentations)
Effectiveness | 6 months
  Total number and type of device related encounters
Effectiveness | 6 months
  Proportion of total device related encounters that are actionable (e.g., changes in programming or treatment)
Connectivity | 6 months
  • Proportion of 24-, 48-, and 72-hour periods with versus without connected wireless monitoring
Quality of Life and Health Status | Baseline, 3 months, and 6 months
  EuroQol 5-dimensional questionnaire, five-level version (EQ-5D-5L) - 5 questions are scored from 1 to 5, with higher scores indicating worse outcomes
Quality of Life and Health Status | Baseline, 3 months, and 6 months
  Cardiac Anxiety Questionnaire (CAQ) - scored from 0 to 72, with a higher score corresponding to higher cardiac anxiety
Quality of Life and Health Status | Baseline, 3 months, and 6 months
  Patient Health Questionnaire depression scale (PHQ-8) - scored from 0 to 24, with a higher score indicating worse symptoms
Quality of Life and Health Status | Baseline, 3 months, and 6 months
  Patient Activation Measure (PAM) - scored from 0 to 100, with a higher score indicating better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided